CLINICAL TRIAL: NCT03839706
Title: Relationship Between 18F-Fluorodeoxyglucose Positron Emission Tomography Magnetic Resonance Imaging Patterns and Circulating Tumor DNA to Predict Hepatocellular Carcinoma Recurrence After Liver Transplantation (PET MRI in HCC)
Brief Title: Relationship Between 18FDG PET/MRI Patterns and ctDNA to Predict HCC Recurrence After Liver Transplantation
Acronym: PETMRIinHCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-6065
Record Dates: First submitted 2019-01-12; First posted 2019-02-15 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET MRI Arm (Experimental): Patient enrolled in the study will have a PET MRI exam scheduled before transplant
  Interventions: Device: PET MRI

INTERVENTIONS:
Device: PET MRI — 18F-Fluorodeoxyglucose Positron Emission Tomography combined with Primovist MRI

SUMMARY:
Liver transplantation is the standard treatment for patients with early-stage Hepatocellular Carcinoma (HCC). Currently, important treatment decisions, like the selection of patients for transplantation, are made on crude, static tumour characteristics such as the size and number of lesions that do not reflect other aspects of tumour biology. To date, pre-transplantation percutaneous biopsy is the best strategy to assess tumoral differentiation and, consequently, tumor biological behavior. Previous studies have demonstrated that 18F-Fluorodeoxyglucose Positron Emission Tomography Magnetic Resonance Imaging (18F-FDG PET/MRI) may have role in assessing the HCC tumoral differentiation and predict survival after LT. The Investigators will assess the accuracy of 18F-FDG PET/MRI as a tool to predict HCC recurrence after liver transplant. To understand the role of 18F-FDG PET/MRI in prediction of HCC's biological behavior and upon recurrence, the investigators will try to assess whether the findings in 18F-FDG PET/MRI can predict HCC poor tumoral differentiation, if the findings in 18F-FDG PET/MRI are related to presence of circulating tumoral DNA in plasma and try to determine the role of 18F-FDG PET/MRI in predicting HCC recurrence after resection. These findings may impact the selection criteria for liver transplantation.

DETAILED DESCRIPTION:
Hepatocellular Carcinoma (HCC) is the third leading cause of death by cancer worldwide, being responsible for nearly 700,000 deaths in 2012. Liver transplantation (LT) provides the best results as a curative treatment for patients with early-stage HCC. Other curative treatment strategies for early stages HCC include resection and ablation. However, the recurrence rates are higher than LT. Due to organ shortage, better criteria for recipient selection are necessary. The first widely accepted criteria for graft allocation in HCC patients is the so-called Milan Criteria (MC): single HCC nodule ≤ 5 cm or 3 nodules all ≤ 3 cm, achieving a 4-y survival of 85%. Recently, MC is seen as too restrictive, its inclusion preventing patients who might have better survival following LT when compared to other therapies. Reluctant to have sizing-only criteria, the University of Toronto, since 2004, has applied the so-called Extended Toronto Criteria (ETC) to LT, which offers transplant to patients with any size and any number of tumors provide they do not have systemic cancer-related symptoms, extrahepatic disease, vascular invasion or poorly differentiated tumors. A recent prospective study conducted at University Health Network (UHN) has shown 5-years survival rates of 68% when ECT are applied. Recent studies have demonstrated the need to use, besides the lesion size, variables which can predict the biological behavior of the tumor.

Currently, important treatment decisions, like the selection of patients for transplantation, are made on crude, static tumour characteristics such as the size and number of lesions, but do not reflect other aspects of tumour biology. To date, pre-transplantation percutaneous biopsy is the best strategy to assess tumor differentiation and, consequently, tumor biological behavior. However, HCC is a very complex disease. Microscopic and molecular analyses have demonstrated a highly heterogeneous degree of cell differentiation. Patients with more than one tumor may have two or three degrees of cell differentiation between the tumors. Even within a single HCC nodule, more than one clonal mutations can be present. To date, there is not a precise method to determinate the degree of differentiation of each patient's disease and percutaneous core biopsy, an invasive method, is the best estimative the investigators can reach.

Since it is impossible to precisely determine the degree of differentiation of HCC with one single tissue sample, the use of imaging becomes necessary. Magnetic resonance imaging (MRI) and enhanced computed tomography (CT) are extensively validated as staging methods for HCC. The use of 18F-Fluorodeoxyglucose (18F-FDG) Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) is still underevaluated in the field of HCC. However, previous studies have demonstrated that 18F-FDG PET/CT may have role in assessing the HCC tumoral differentiation and predict survival after LT. There is no investigation on use of 18F-FDG PET/MRI as a tool to predict biological behavior in HCC.

Recently, the Pugh Lab has developed a circulating tumor DNA (ctDNA) sequencing assay that combines a hybrid-capture method with a novel bioinformatics algorithm to enable full-length sequence analysis of all exons in genes of interest or any other arbitrary genomic region, rather than mutation hotspots13. With the availability of these technologies in our group, the investigators next sought to determine whether these methods were applicable to HCC patients, gathering two innovative tools in transplant patients' care.

ELIGIBILITY:
Inclusion Criteria:

* Histological or radiological diagnosis of HCC (AASLD guidelines)
* Listed for LT at UHN
* Enrolled in ctDNA study (15-5925)
* Able to undergo PET and MRI examination,
* Willingness and ability of patient to provide signed voluntary informed consent.
* Adults (age ≥ 18-years old)

Exclusion Criteria:

* Any contraindication to undergoing venipuncture.
* Patients with previous history of cancer diagnosed and/or treated within last 5 years, with the exception of non-melanomatous skin cancers and intraepithelial cancers such as cervical intraepithelial neoplasia that were properly treated, are not eligible.
* Inability to lie supine for at least 30 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
18F-FDG PET/MRI results can identify aggressive HCC behavior and recurrence post transplant | 3 years
  PET scan results will be compared with pathology at the time of transplant. Patients will be followed-up 2 years post transplant for recurrence. PET scan results will be compared for Recurrent/non-recurrent patients.

SECONDARY OUTCOMES:
18F-FDG PET/MRI can predict HCC's poor tumoral differentiation | 3 years
  PET/MRI reports will be compared with pathology at the time of transplant.
18F-FDG PET/MRI are related to presence of circulating tumor DNA in plasma | 3 years
  18F-FDG PET/MRI scan results will be compared with levels of ctDNA identified in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada